CLINICAL TRIAL: NCT02521935
Title: Conventionally vs. Digitally Fabricated Complete Dentures: Clinical Treatment Outcome Differences
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI is deceased, decision was made to withdraw.
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Global Dental Science, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14-1811
Record Dates: First submitted 2015-07-16; First posted 2015-08-13 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Mouth, Edentulous
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Complete traditional dentures (Active Comparator): Complete maxillary/mandible dentures made in the traditional manner.
  Interventions: Device: Complete traditional dentures
- Complete CADCAM dentures (Active Comparator): Complete maxillary/mandible dentures made with CADCAM (computer-aided design/computer-aided manufacturing) technology
  Interventions: Device: Complete CADCAM dentures

INTERVENTIONS:
Device: Complete traditional dentures — Arm 1-Standard Treatment Sequence for Traditional Removable Dentures in a Dental School Clinic (9 Appointments):
  Appointment 1: Examination & diagnosis & initial impressions.
  Appointment 2: Secondary impressions.
  Appointment 3: Secondary or definitive impressions (Often 2 appointments are needed to border mold and impression)
  Appointment 4: Maxillo-mandibular jaw relation records (both centric and vertical relation). Tooth selection.
  Appointment 5: Wax-trial denture try-in.
  Appointment 6: Insertion and instructions for care of definitive prostheses.
  Appointments 7-9 Post adjustments
  Other Names: complete conventional dentures
  Arms: Complete traditional dentures
Device: Complete CADCAM dentures — Arm 2-Standard Treatment Sequence for Digital Dentures in a Dental School Clinic (5 appointments):
  Appointment 1: Exam, diagnosis, & tray selection (begin impressions)
  Appointment 2: Definitive impressions and Maxillomandibula relations
  Appointment 3: Wax-trial arrangement
  Appointment 4: Insertion and instructions for care of definitive prosthesis
  Appointment 5: Post adjustment/s (Less post insertion adjustments are anticipated due to CADCAM milling of the denture base and less polymerization shrinkage
  Other Names: complete digital dentures
  Arms: Complete CADCAM dentures

SUMMARY:
Purpose: To compare complete denture outcomes between conventional and digital denture fabrication processes.

Participants: Sixteen edentulous adult patients in the University of North Carolina School of Dentistry Student Clinic who are seeking removable complete dentures.

Procedures (methods): Two complete sets of dentures will be fabricated for each subject: one using the conventional process (A) and the other using a digital process (B). Variability will be assessed by the research team, the treating dental students, an independent prosthodontist, and the patients through quantitative measures. Case selection and results analysis will be evaluated with recognition of the Prosthodontic Diagnostic Index.

DETAILED DESCRIPTION:
Rationale for Study Design An AB/BA (conventional=A, digital=B) crossover design with no wash-out period is flawed for this study, and its weakness is the potential for a carryover effect (benefits or risks associated with treatment A carry over to treatment B). A wash-out period is not feasible for this study because it would require the patient-subjects to suspend use of their dentures for the duration of the wash-out period.

The Investigators have decided to conduct the study using the ABB/BAA crossover design, which does not require a wash-out period and will permit testing and discounting of a possible carryover effect. In addition, this design is more appropriate for a small sample size than the AB/BA design.

The investigators are adding to the scant literature on digital dentures, information that has never before been studied - the retention, aesthetics, and stability of digital dentures compared to conventional dentures. Additionally, the investigators will have longitudinal data on these characteristics regarding digital dentures.

If the Functional Assessment of Dentures (FAD) and the patient evaluation show positive results for the digital dentures, this could lead to increased use of the Computer -Aided Design/ Computer -Aided Manufacturing (CADCAM) fabrication method which, in turn, would allow greater numbers of people to benefit from the advantages of the digital dentures as described earlier in this application (e.g., a better fit, fewer visits with less time in the chair, less biofilm formation, etc.)

ELIGIBILITY:
Inclusion Criteria:

1. UNC School of Dentistry Student Clinic patients requiring maxillary and mandibular complete dentures
2. Ages 18 to 99, inclusive
3. Able to read, speak, and understand English
4. Without natural tooth or implant supported overdentures
5. Edentulous in both jaws for at least 6 months
6. Any Prosthodontic Diagnostic Index (PDI) type with a preference given to Types 1-3

Exclusion Criteria:

1. Non-registered patient in UNC School of Dentistry student clinics
2. Patient not able or unwilling to give consent
3. Subject had extractions within last 6 months

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2018-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
the overall comparison of functional assessment of digitally fabricated dentures to traditionally fabricated dentures | 2 years
  evaluate functional assessment of digitally fabricated dentures to traditionally fabricated dentures (FAD= Functional Assessment of Dentures)

SECONDARY OUTCOMES:
comparison of functional assessment of digitally fabricated dentures to traditionally fabricated dentures | baseline = 4 weeks
  evaluate functional assessment of digitally fabricated dentures to traditionally fabricated dentures (FAD= Functional Assessment of Dentures)
comparison of functional assessment of digitally fabricated dentures to traditionally fabricated dentures | 3 months
  evaluate functional assessment of digitally fabricated dentures to traditionally fabricated dentures (FAD)
comparison of functional assessment of digitally fabricated dentures to traditionally fabricated dentures | 6 months
  evaluate functional assessment of digitally fabricated dentures to traditionally fabricated dentures (FAD)
comparison of functional assessment of digitally fabricated dentures to traditionally fabricated dentures | 1 year
  evaluate functional assessment of digitally fabricated dentures to traditionally fabricated dentures (FAD)
comparison of patient satisfaction between digital dentures and traditional dentures | baseline = 4 weeks
  patient satisfaction survey consisting of 12 items organized into 5 subscales (not at all satisfied, not very satisfied, reasonably satisfied, very satisfied, totally satisfied) and responses are based on a Likert scale
comparison of patient satisfaction between digital dentures and traditional dentures | 3 months
  patient satisfaction survey consisting of 12 items organized into 5 subscales (not at all satisfied, not very satisfied, reasonably satisfied, very satisfied, totally satisfied) and responses are based on a Likert scale
comparison of patient satisfaction between digital dentures and traditional dentures | 6 months
  patient satisfaction survey consisting of 12 items organized into 5 subscales (not at all satisfied, not very satisfied, reasonably satisfied, very satisfied, totally satisfied) and responses are based on a Likert scale
comparison of patient satisfaction between digital dentures and traditional dentures | 1 year
  patient satisfaction survey consisting of 12 items organized into 5 subscales (not at all satisfied, not very satisfied, reasonably satisfied, very satisfied, totally satisfied) and responses are based on a Likert scale
comparison of patient satisfaction between digital dentures and traditional dentures | 2 year
  patient satisfaction survey consisting of 12 items organized into 5 subscales (not at all satisfied, not very satisfied, reasonably satisfied, very satisfied, totally satisfied) and responses are based on a Likert scale
bite force comparison between digital dentures and traditional dentures | baseline = 4 weeks
  using gnathometer assessment, investigators will record the force (on a 0-10 scale) during dislodgement
bite force comparison between digital dentures and traditional dentures | 3 months
  using gnathometer assessment, investigators will record the force (on a 0-10 scale) during dislodgement
bite force comparison between digital dentures and traditional dentures | 6 months
  using gnathometer assessment, investigators will record the force (on a 0-10 scale) during dislodgement
bite force comparison between digital dentures and traditional dentures | 1 year
  using gnathometer assessment, investigators will record the force (on a 0-10 scale) during dislodgement
bite force comparison between digital dentures and traditional dentures | 2 year
  using gnathometer assessment, investigators will record the force (on a 0-10 scale) during dislodgement

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Wright, DDS FACP, Principal Investigator — Professor and Chair, Dept. of Prosthodontics UNC School of Dentistry
Locations (1):
- University of North Carolina School of Dentistry Student Clinics, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCord JF. Contemporary techniques for denture fabrication. J Prosthodont. 2009 Feb;18(2):106-11. doi: 10.1111/j.1532-849X.2009.00439.x. PMID 19254299
- [Background] Goodacre CJ, Garbacea A, Naylor WP, Daher T, Marchack CB, Lowry J. CAD/CAM fabricated complete dentures: concepts and clinical methods of obtaining required morphological data. J Prosthet Dent. 2012 Jan;107(1):34-46. doi: 10.1016/S0022-3913(12)60015-8. PMID 22230914
- [Background] Lee WS, Kim WC, Kim HY, Kim WT, Kim JH. Evaluation of different approaches for using a laser scanner in digitization of dental impressions. J Adv Prosthodont. 2014 Feb;6(1):22-9. doi: 10.4047/jap.2014.6.1.22. Epub 2014 Feb 14. PMID 24605202
- [Background] Kattadiyil MT, Goodacre CJ, Baba NZ. CAD/CAM complete dentures: a review of two commercial fabrication systems. J Calif Dent Assoc. 2013 Jun;41(6):407-16. PMID 23875432
- [Background] Bidra AS, Taylor TD, Agar JR. Computer-aided technology for fabricating complete dentures: systematic review of historical background, current status, and future perspectives. J Prosthet Dent. 2013 Jun;109(6):361-6. doi: 10.1016/S0022-3913(13)60318-2. PMID 23763779
- [Background] Darvell BW, Clark RK. The physical mechanisms of complete denture retention. Br Dent J. 2000 Sep 9;189(5):248-52. doi: 10.1038/sj.bdj.4800734. PMID 11048392
- [Background] Parvizi A, Lindquist T, Schneider R, Williamson D, Boyer D, Dawson DV. Comparison of the dimensional accuracy of injection-molded denture base materials to that of conventional pressure-pack acrylic resin. J Prosthodont. 2004 Jun;13(2):83-9. doi: 10.1111/j.1532-849X.2004.04014.x. PMID 15210003
- [Background] Infante L, Yilmaz B, McGlumphy E, Finger I. Fabricating complete dentures with CAD/CAM technology. J Prosthet Dent. 2014 May;111(5):351-5. doi: 10.1016/j.prosdent.2013.10.014. Epub 2014 Jan 23. PMID 24461946
- [Background] Alfadda SA. The relationship between various parameters of complete denture quality and patients' satisfaction. J Am Dent Assoc. 2014 Sep;145(9):941-8. doi: 10.14219/jada.2013.48. PMID 25170001
- [Background] Allen PF, McMillan AS, Walshaw D. A patient-based assessment of implant-stabilized and conventional complete dentures. J Prosthet Dent. 2001 Feb;85(2):141-7. doi: 10.1067/mpr.2001.113214. PMID 11208203
- [Background] Anastassiadou V, Naka O, Heath MR, Kapari D. Validation of indices for functional assessment of dentures. Gerodontology. 2002 Jul;19(1):46-52. doi: 10.1111/j.1741-2358.2002.00046.x. PMID 12164239
- [Background] Corrigan PJ, Basker RM, Farrin AJ, Mulley GP, Heath MR. The development of a method for functional assessment of dentures. Gerodontology. 2002 Jul;19(1):41-5. doi: 10.1111/j.1741-2358.2002.00041.x. PMID 12164238
- [Background] Fenlon MR, Sherriff M, Walter JD. An investigation of factors influencing patients' use of new complete dentures using structural equation modelling techniques. Community Dent Oral Epidemiol. 2000 Apr;28(2):133-40. doi: 10.1034/j.1600-0528.2000.028002133.x. PMID 10730722
- [Background] Sato Y, Hamada S, Akagawa Y, Tsuga K. A method for quantifying overall satisfaction of complete denture patients. J Oral Rehabil. 2000 Nov;27(11):952-7. doi: 10.1046/j.1365-2842.2000.00579.x. PMID 11106986
- [Background] Sato Y, Tsuga K, Akagawa Y, Tenma H. A method for quantifying complete denture quality. J Prosthet Dent. 1998 Jul;80(1):52-7. doi: 10.1016/s0022-3913(98)70091-5. PMID 9656178
- [Background] WOELFEL JB, PAFFENBARGER GC, SWEENEY WT. CLINICAL EVALUATION OF COMPLETE DENTURES MADE OF 11 DIFFERENT TYPES OF DENTURE BASE MATERIALS. J Am Dent Assoc. 1965 May;70:1170-88. doi: 10.14219/jada.archive.1965.0208. No abstract available. PMID 14284642